CLINICAL TRIAL: NCT06429254
Title: Effect of Emotional Freedom Techniques on Pelvic Pain and Quality of Life in Women With Endometriosis: A Randomized Controlled Study
Brief Title: The Effect of Emotional Freedom Techniques on Pelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Ayse Cuvadar, Assistant Professor, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 01/05
Record Dates: First submitted 2024-04-27; First posted 2024-05-24 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Woman; Pelvic Pain
Keywords: Pelvic pain; Woman; quality of life
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotional Freedom Techniques group (Experimental): First, the Personal Information Form, Visual Analogue Scale, and Quality of Life Scale will be administered as pre-tests to the EFT group. A high score obtained from the quality of life scale indicates a high quality of life.
  After the pre-tests, the first EFT session will be conducted. A second EFT session will take place 30 days later, followed by post-tests. During this period, affirmations will be provided as needed based on individual difficulties, perspectives, support systems, past traumas, and emotional blockages experienced by the woman. Each session is planned to last approximately 45 minutes to 1 hour.
  Procedure: Administering pre-tests followed by the first EFT session. Procedure: After 30 days, conducting post-tests followed by the second EFT session.
  Procedure: After another 30 days, only post-tests will be conducted.
  Interventions: Other: Experimental group
- Control group (No Intervention): After obtaining consent from the women included in the group, pre-tests will be conducted followed by breathing exercises. A program will be tailored according to the suitability of the women. Once an appropriate environment is provided for meeting with the women, information about the study will be provided. Pain coping methods will be explained, and breathing exercises will be taught. The exercises will commence when the woman feels ready. The breathing exercises typically last around 15-20 minutes.
  With a plan for a total of 8 breathing exercises to be conducted over four weeks, consisting of 2 sessions per week, they will be scheduled to coincide with the EFT group, with sessions held every 5 days.

INTERVENTIONS:
Other: Experimental group — Life Scale will be administered as pre-tests to the EFT group. After the pre-tests, the first EFT session will be conducted. A second EFT session will take place 30 days later, followed by post-tests. During this period, affirmations will be provided as needed based on individual difficulties, perspectives, support systems, past traumas, and emotional blockages experienced by the woman. Each session is planned to last approximately 45 minutes to 1 hour.
  Other Names: EFT group
  Arms: Emotional Freedom Techniques group

SUMMARY:
Pelvic pain caused by endometriosis is a common symptom and reduces women's quality of life.

EFT is a method that can be preferred in pelvic pain due to its ease of use and low cost.

Raising women's awareness for EFT

DETAILED DESCRIPTION:
Pelvic pain caused by endometriosis is a common symptom and reduces women's quality of life. EFT has become widely used in medical and psychological treatment settings in recent years.It is also used as a self-help technique by millions of people every year.EFT is a method that can be preferred in pelvic pain due to its ease of use and low cost.

ELIGIBILITY:
Inclusion Criteria:

1. Being diagnosed with endometriosis
2. Experiencing pelvic pain
3. Being between the ages of 18-49
4. Those whose symptom complaints are 5 or above on the visual analogue scale

Exclusion Criteria:

1. Patients with known systemic diseases (e.g. hypertension, diabetes, coronary, kidney and liver diseases);
2. Patients with known malignancy;
3. Women in menopause;
4. Having any obstacle to communication

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women
Enrollment: 64 (Actual)
Dates: Start 2024-05-24 (Actual); Primary Completion 2024-10-27 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Examining the Effect of Emotional Freedom Technique on Pelvic Pain in Endometriosis | 2 months; participants will receive 2 EFT sessions, one session per month. Pain and quality of life will be assessed at baseline and after 2 months.
  Primary Outcome Measures: Pain measured using the Visual Analog Scale (VAS); higher scores indicate greater pain.
  Secondary Outcome Measures: Quality of life measured using the SF-36; higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya University, Edirne, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No